CLINICAL TRIAL: NCT02386566
Title: A Prospective, Multicenter, Observational Study to Assess the Correlation of EDSS With Quality of Life in MS Patients Treated With Natalizumab
Brief Title: Observational Study to Assess the Correlation of EDSS With Quality of Life in MS Participants Treated With Natalizumab
Acronym: PROTYS
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: CHE-TYS-12-10341
Record Dates: First submitted 2015-02-06; First posted 2015-03-12 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- natalizumab: natalizumab 300 mg intravenous (IV) every 4 weeks; according to the approved product label of Tysabri in Switzerland
  Interventions: Drug: natalizumab

INTERVENTIONS:
Drug: natalizumab — As described in the treatment arm
  Other Names: Tysabri; BG00002

SUMMARY:
The primary objective of the study is to determine the association between prospectively measured disability (Expanded Disability Status Scale [EDSS]) with quality of life (Multiple Sclerosis International Quality of Life Questionnaire [MusiQoL]) at 3-month intervals up to 1 year in a real life setting of multiple sclerosis (MS) patients treated with natalizumab. The secondary objectives of this study are as follows: To evaluate the cumulative probability of sustained EDSS changes at 1 year following natalizumab treatment initiation; To evaluate the association between disability (EDSS), fatigue (Fatigue Scale of Motor and Cognitive Function [FSMC]), sexual dysfunction (Multiple Sclerosis Intimacy and Sexuality Questionnaire-19 [MSISQ-19]), depression (Beck Depression Inventory-Fast Screen [BDI-FS]) and neurocognitive function (Symbol Digit Modalities Test [SDMT]) with EuroQol-5D Questionnaire (EQ-5D) at 3 to 6-months intervals up to 1 year after initiation of natalizumab treatment; To assess the relationship between clinical disease-free status (no EDSS increase of 1.0 and no relapse) and MusiQoL at 1 year following natalizumab treatment initiation; To record the number of clinical relapses and relapses requiring steroid treatment at 3-months intervals up to 1 year after initiation of natalizumab treatment; To describe changes in work impairment (Work Productivity and Activity Impairment in MS [WPAI-MS]) at 3-months intervals up to 1 year after initiation of natalizumab treatment; To describe any change in the percentage of disability pension and occupation after 1 year of natalizumab treatment; To record the incidence and number of Serious Adverse Events (SAE) and Suspected Unexpected Serious Adverse Reactions (SUSAR) throughout the study

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects that have a confirmed diagnosis of RRMS, as per the 2010 revised McDonald criteria
* Subjects satisfying the therapeutic indication of natalizumab, as described in the local product label and confirmed by the Investigator. (Patients with previous treatment with natalizumab are also considered to be eligible only if the last natalizumab infusion was at least 1 year before the screening visit of this study)
* Decision for a treatment with natalizumab has been made before screening
* Patients with an EDSS score of 2.0-5.5 (both limits inclusive)

Key Exclusion Criteria:

* Patients with a diagnosed co-existing brain pathology other than MS, which in the judgement of the investigator impacts the value of EDSS or QoL.
* Pure spinal manifestation of demyelination
* Diagnosis of primary or secondary progressive MS
* Any change in concomitant medication known to affect cognition or bladder function
* A history of severe depressive disorder and/or suicidality, seizure, drug or alcohol abuse, as assessed by the Investigator

NOTE: Other Protocol Defined Inclusion/ Exclusion Criteria May Apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with relapsing remitting multiple sclerosis (RRMS) that have been prescribed natalizumab under standard clinical care.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2015-03-20 (Actual); Primary Completion 2018-01-28 (Actual); Study Completion 2018-01-28 (Actual)

PRIMARY OUTCOMES:
Compare EDSS change categories with changes in MusiQoL | At 1 year after initiating natalizumab treatment
  The EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. Scoring is based on measures of impairment in eight functional systems on examination by a neurologist. The MusiQOL is a multidimensional Health Related Quality of Life (HRQoL) instrument that provides information based on the views and perceptions of the participants.

SECONDARY OUTCOMES:
Cumulative probabilities of sustained improvement and progression in neurological disability | At 1 year after initiating natalizumab treatment
Compare clinical disease-free status (no sustained EDSS increase of 1.0 and no relapse) with MusiQoL | Up to 1 year after initiating natalizumab treatment
Compare EDSS change categories with EQ-5D | Up to 1 year after initiating natalizumab treatment
  The EQ-5D is a two-part instrument that consists of the following administered together: 1) EQ-5D-5L- The descriptive system comprises the same 5 dimensions as the EQ-5D-3L (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each dimension now has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. EQ-VAS describes the respondent's self-rated health on a vertical visual analog scale (VAS).
Compare FSMC score with EQ-5D | Up to 1 year after initiating natalizumab treatment
  FSMC provides differential quantification and graduation of cognitive and motor fatigue. The total score ranges from 0 to 100 with higher scores indicating more fatigue.
Compare MSISQ-19 scores with EQ-5D | Up to 1 year after initiating natalizumab treatment
  MSIS-Q is a 19-question survey to assess sexual QoL in MS patients. The scoring is based on a scale ranging from 1 (never interfered with my sexual activity or satisfaction) to 5 (always interfered with my sexual activity or satisfaction).
Comparison of BDI-FS with EQ-5D | Up to 1 year after initiating natalizumab treatment
  The Beck Depression Inventory (BDI) as measured by the BDI-FS is a 7-item multiple-choice self-report inventory for measuring the severity of depression in MS.
Compare SDMT scores with EQ-5D | Up to 1 year after initiating natalizumab treatment
  SDMT is a screening test for cognitive impairment. It assesses key neurocognitive functions that underlie many substitution tasks, including attention, visual scanning, and motor speed. SDMT scores are highly correlated to Magnetic Resonance Imaging (MRI) derived measures of disease burden and disability progression in MS patients.
Rates of clinical relapses and relapses requiring steroid treatment | Up to 1 year after initiating natalizumab treatment
Changes in the WPAI questionnaire | Up to 1 year after initiating natalizumab treatment
  The WPAI questionnaire is a validated instrument to measure impairments in work and activities. The WPAI yields four types of scores: 1. Absenteeism (work time missed) 2. Presenteesism (impairment at work / reduced on-the-job effectiveness) 3. Work productivity loss (overall work impairment / absenteeism plus presenteeism) 4. Activity Impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Change in kind and percentage of occupation due to MS | At 1 year after initiating natalizumab treatment
Change in the percentage of disability pension | At 1 year after initiating natalizumab treatment
Incidence and number of SAEs and SUSARs | Up to 1 year after initiating natalizumab treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (7):
- Switzerland (7):
  - Research Site, Aarau
  - Research Site, Basel
  - Research Site, Bern
  - Research site - private practice, Lucerne
  - Research Site, Lugano
  - Research Site, Wohlen
  - Research Site, Zurich

REFERENCES:
- [Derived] Achtnichts L, Zecca C, Findling O, Kamm CP, Mueller S, Kuhle J, Lutterotti A, Gobbi C, Viviani C, Villiger-Borter E, Nedeltchev K. Correlation of disability with quality of life in patients with multiple sclerosis treated with natalizumab: primary results and post hoc analysis of the TYSabri ImPROvement study (PROTYS). BMJ Neurol Open. 2023 Jan 26;5(1):e000304. doi: 10.1136/bmjno-2022-000304. eCollection 2023. PMID 36727105